CLINICAL TRIAL: NCT05347368
Title: Effects of Primal Reflex Release Technique on Pain, Disability and Flexibility in Patients With Chronic Non-specific Low Back Pain
Brief Title: Effects of Primal Reflex Release Technique in Chronic Non-specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0131 Aleena
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: Low Back pain; Disability; Flexibility; Primal Reflex; Autonomic Nervous system
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (conventional therapy) (Other)
  Interventions: Other: Control group (conventional therapy)
- Primal Reflex release Technique (Experimental)
  Interventions: Other: Control group (conventional therapy); Other: Primal Reflex release Technique

INTERVENTIONS:
Other: Control group (conventional therapy) — Physical therapy will be performed using physical agent modality that include hot pack (15 min), and therapeutic exercises (5 repetition per set, 2 sets each session) therapeutic exercises include spinal extension exercise, prone hip extension exercise, posterior pelvic tilt, cat-camel exercise
Other: Primal Reflex release Technique — The SI/Lumbar release Iliopsoas release Piriformis release Hamstring release Gastrocnemius release
  Arms: Primal Reflex release Technique

SUMMARY:
Low back pain is a major disorder which occurs from chronic over use and injury to lumbar musculoskeletal system. Sometimes the source of pain is non-specific leading to pain and spasm due to muscle imbalance. Primal reflex release technique is a novel concept to decrease pain and muscle spasm by resetting reflexes using reciprocal inhibition following the concept of rebooting the Autonomic nervous system. This study aims to determine the effects of primal reflex release technique on pain, flexibility and disability in chronic nonspecific low back pain patients.

This study will be a Randomized Controlled trial and will be conducted at Arif Memorial Hospital in Lahore. A sample size of Total 32 patients will be taken in this study using consecutive sampling technique. Patients will be randomly assigned into two groups.

Group A will be treated by conventional therapy and Group B will be treated by conventional therapy and primal reflex release technique. Numeric Pain Rating Scale and Ronald Morris Disability Questionnaire will be used to evaluate pain and disability respectively. Flexibility of low back, Iliopsoas, hamstring, Piriformis and gastrocnemius will be measured by schober's test, modified Thomas test, Active knee extension test, FAIR test and active dorsiflexion, respectively. The evaluation will be on day 1 as pretreatment values and at 2nd and 4th week as post treatment values respectively. The collected data will be analyzed on SPSS - 25.

ELIGIBILITY:
Inclusion Criteria:

Age 25-45

* Both males and females
* Lower cross syndrome diagnosed by straight leg raise, modified Thomas test, piriformis stretch test.
* History of LBP for more than 6 weeks before the study, or had on-and-off pain having suffered at least 3 episodes of LBP during the year before the study, each lasting more than a year
* The diagnosis confirmed on the presence of -pain experienced between the costal margins and the inferior gluteal folds which is influenced by physical activities and postures, usually accompanied by painful limitation of motion‖

Exclusion Criteria:

No recent history of injury to lower limb

* No experience with surgical treatments for disc herniation, spina bifida, or spinal stenosis,
* No nerve root compression or no neurological problems.
* SIJ compression test positive

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 week
  Patient level of pain will be evaluated by using the NPRS (0-10 with 0 representing -no pain‖ and 10 the -worst pain‖). Clinometric properties of the NPRS are well established .The NPRS minimal clinically important difference (MCID) is 2 points
Ronald Morris Disability Questionnaire | 4 weeks
  To measure the level of disability caused by CLBP, we will use the Ronald Morris disability questionnaire RMDQ (0-24, with 0 representing no disability and 24 the most disability), which has good internal consistency (Cronbach's alpha =0.83) and test-retest reliability (interclass correlation coefficient= 0.87). Its MCID varies between 1-2 points in patients with minimal disability and 7-8 points in patients with severe disability
Schober's Test | 4 weeks
  The schober's test will be used to assess flexibility in the lower back. Schober's test will be applied to assess spinal mobility, with participants standing at maximal spinal flexion. The reference points will be near the fifth lumbar vertebra (between the posterior superior iliac spines) and 10 cm above this point. The test will be considered normal when there is difference of five or more centimeters between standing upright and at maximal spinal flexion
Ankle Knee Extension Test | 4 weeks
  The Ankle knee extension test (TTT) will be used to measure hamstring muscle flexibility. In this test, each subject will be in supine position, with a small pillow beneath his head and neck. The knee flexion axis will be marked by a pen and from this point, a line will be drawn to the greater trochanter of the femur and one other line to the external malleolus of the ankle. These lines will be used to measure knee joint angles. The goniometer axis will be on the knee axis and its arm will be along the line drawn on the thigh and the other arm will be along the line drawn on the leg. The subject will be asked to do the active knee extension slowly within 3 s as far as he/she could while the ankle remains in a neutral position. Then, when the active knee extension movement will complete and the subject will attempt to keep this situation for a second, the angle indicated by the goniometer will be extension angle of the knee joint
Modified Thomas Test | 4 weeks
  The modified Thomas test (MTT) will be used to measure Iliopsoas muscle flexibility
FAIR (Flexion Adduction internal rotation) Test | 4 weeks
  The flexion adduction internal rotation test (FAIRT) will be used to measure Piriformis muscle flexibility
Active Ankle Dorsiflexion Test | 4 weeks
  The Active Ankle Dorsiflexion will be used to measure gastrocnemius flexibility.

SECONDARY OUTCOMES:
Patient Global Impression Of Change | 4 weeks
  The perception of improvement after treatment will be assessed by the patient global impression of change PGIC (range 0-7) (23). This scale is valid and recommended for patients with chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Arif Memorial Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghorbanpour A, Azghani MR, Taghipour M, Salahzadeh Z, Ghaderi F, Oskouei AE. Effects of McGill stabilization exercises and conventional physiotherapy on pain, functional disability and active back range of motion in patients with chronic non-specific low back pain. J Phys Ther Sci. 2018 Apr;30(4):481-485. doi: 10.1589/jpts.30.481. Epub 2018 Apr 13. PMID 29706690
- [Background] Rooh Ul Muazzam M, Abbas S, Abbas S, Rafi MA. Frequency of low back pain in young adults and its relationship with different mattresses. J Pak Med Assoc. 2021 Sep;71(9):2177-2180. doi: 10.47391/JPMA.03-494. PMID 34580510
- [Background] Ijaz M, Akram M, Ahmad SR, Mirza K, Ali Nadeem F, Thygerson SM. Risk Factors Associated with the Prevalence of Upper and Lower Back Pain in Male Underground Coal Miners in Punjab, Pakistan. Int J Environ Res Public Health. 2020 Jun 9;17(11):4102. doi: 10.3390/ijerph17114102. PMID 32526830
- [Background] Alsufiany MB, Lohman EB, Daher NS, Gang GR, Shallan AI, Jaber HM. Non-specific chronic low back pain and physical activity: A comparison of postural control and hip muscle isometric strength: A cross-sectional study. Medicine (Baltimore). 2020 Jan;99(5):e18544. doi: 10.1097/MD.0000000000018544. PMID 32000363
- [Background] Chatchawan U, Jupamatangb U, Chanchitc S, Puntumetakul R, Donpunha W, Yamauchi J. Immediate effects of dynamic sitting exercise on the lower back mobility of sedentary young adults. J Phys Ther Sci. 2015 Nov;27(11):3359-63. doi: 10.1589/jpts.27.3359. Epub 2015 Nov 30. PMID 26696698
- [Background] Sahin N, Karahan AY, Albayrak I. Effectiveness of physical therapy and exercise on pain and functional status in patients with chronic low back pain: a randomized-controlled trial. Turk J Phys Med Rehabil. 2017 Aug 9;64(1):52-58. doi: 10.5606/tftrd.2018.1238. eCollection 2018 Mar. PMID 31453489
- [Background] Kim B, Yim J. Core Stability and Hip Exercises Improve Physical Function and Activity in Patients with Non-Specific Low Back Pain: A Randomized Controlled Trial. Tohoku J Exp Med. 2020 Jul;251(3):193-206. doi: 10.1620/tjem.251.193. PMID 32669487
- [Background] Albertin ES, Walters M, May J, Baker RT, Nasypany A, Cheatham S. AN EXPLORATORY CASE SERIES ANALYSIS OF THE USE OF PRIMAL REFLEX RELEASE TECHNIQUE TO IMPROVE SIGNS AND SYMPTOMS OF HAMSTRING STRAIN. Int J Sports Phys Ther. 2020 Apr;15(2):263-273. PMID 32269860
- [Background] Behennah J, Conway R, Fisher J, Osborne N, Steele J. The relationship between balance performance, lumbar extension strength, trunk extension endurance, and pain in participants with chronic low back pain, and those without. Clin Biomech (Bristol). 2018 Mar;53:22-30. doi: 10.1016/j.clinbiomech.2018.01.023. Epub 2018 Jan 31. PMID 29407352
- [Background] O'Keeffe M, O'Sullivan P, Purtill H, Bargary N, O'Sullivan K. Cognitive functional therapy compared with a group-based exercise and education intervention for chronic low back pain: a multicentre randomised controlled trial (RCT). Br J Sports Med. 2020 Jul;54(13):782-789. doi: 10.1136/bjsports-2019-100780. Epub 2019 Oct 19. PMID 31630089